CLINICAL TRIAL: NCT04402060
Title: A Randomized, Double-Blinded, Vehicle-Controlled, Multicenter, Parallel-Group Study of APL-9 in Mild to Moderate Acute Respiratory Distress Syndrome Due to COVID-19
Brief Title: A Study of APL-9 in Adults With Mild to Moderate ARDS Due to COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APL9-COV-201
Record Dates: First submitted 2020-05-22; First posted 2020-05-26 (Actual); Results first posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: COVID; Covid-19; Coronavirus; Coronavirus Infection; Severe Acute Respiratory Syndrome; Severe Acute Respiratory Syndrome Coronavirus 2; Sars-CoV2; Ards; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome; Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 180 mg APL-9 IV plus SOC (Experimental)
  Interventions: Drug: APL-9
- Isotonic saline plus SOC (Placebo Comparator)
  Interventions: Other: Vehicle Control

INTERVENTIONS:
Drug: APL-9 — Complement (C3) Inhibitor
  Arms: 180 mg APL-9 IV plus SOC
Other: Vehicle Control — Normal saline of equal volume to active arm
  Arms: Isotonic saline plus SOC

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of APL-9 in adults with mild to moderate ARDS (acute respiratory distress syndrome) caused by COVID-19 who are hospitalized and require supplemental oxygen therapy with or without mechanical ventilation.

It is thought that COVID-19 activates the complement system, part of the immune system that responds to infection or tissue damage, and increases inflammation in the lungs. APL-9 has been designed to inhibit or block activation of part of the complement pathway, and potentially reduce inflammation in the lungs.

Part 1 of the study is open-label to evaluate safety; all participants will receive APL-9 plus standard of care. Part 2 of the study is double-blind, randomized; participants will receive either APL-9 or the vehicle-control plus standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age at time of informed consent
* Diagnosis of active SARS CoV 2 infection using viral RNA or viral antigen within 7 days of screening
* Respiratory failure requiring oxygen supplementation or either invasive or noninvasive mechanical ventilation with PaO2/FiO2 ratio >100 mm Hg. Respiratory failure cannot be fully explained by cardiac failure or fluid overload.

Exclusion Criteria:

* Treatment with immune checkpoint inhibitors, or other immunomodulators within 3 months prior to study enrollment (however, treatment with convalescent plasma, steroids, IL-6 inhibitors, and antiviral agents is NOT excluded)
* Active bacterial, fungal, or parasitic infection
* History of neuromuscular degenerative disease (eg, amyotrophic lateral sclerosis, Duchenne muscular dystrophy, or multiple sclerosis)
* Current participation in an interventional clincial trial
* Subjects who have, at screening, been on mechanical ventilation for >7 days Have evidence of kidney and liver failure at screening
* Have a hereditary complement deficiency
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-02-13 (Actual); Study Completion 2021-02-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (16):
  - University of California at San Francisco - Fresno, Fresno, California
  - California Pacific Medical Center, San Francisco, California
  - Baptist Medical Center Beaches, Jacksonville Beach, Florida
  - Westchester General Hospital, Miami, Florida
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran Health Physicians, Fort Wayne, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Norton Women's and Children's Hospital, Louisville, Kentucky
  - Norton Audobon Hospital, Louisville, Kentucky
  - Cambridge Medical Trials, Alexandria, Louisiana
  - Ascension Providence Hospital, Southfield, Michigan
  - Rutgers University - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University at Buffalo, Buffalo, New York
  - Columbia University, New York, New York
  - Texas A&M College of Medicine - Scott and White, Temple, Texas
- Brazil (8):
  - Hospital Angelina Caron, Campina Grande do Sul, Paraná
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - UPECLIN - Unidade de Pesquisa Clínica da Faculdade de Medicina de Botucatu - FMB/UNESP, Botucatu, São Paulo
  - Hospital Estadual Mario Covas, Santo André, São Paulo
  - CEMEC - Centro Multidisciplinar de Estudos Clinicos LTDA EPP, São Bernardo do Campo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, vehicle-controlled, multicenter, parallel-group Phase 1/2 study (with an initial open-label period) evaluating the safety and efficacy of APL-9 versus (vs) vehicle control as an add-on therapy to standard of care (SoC) in subjects who had respiratory failure, including mild to moderate acute respiratory distress syndrome (ARDS) due to coronavirus disease 2019 (COVID-19).
Pre-assignment Details: The study was conducted in 2 parts: Subjects in Part 1 received open-label APL-9 from Day 1 through Day 7 or resolution of ARDS. Subjects in Part 2 were randomly assigned 1:1 to blinded treatment with either APL-9 or vehicle control from Day 1 through Day 7 or up to and including Day 21, discontinuation of respiratory support or hospital discharge, whichever occurred latest. Extended treatment beyond Day 7 in Part 2 required certain criteria to be met and was at discretion of the Investigator.
Groups:
- Part 1: APL-9: Subjects received an initial intravenous (IV) infusion of 180 milligram (mg) APL-9 in 50 milliliter (mL) of saline once over a 10-minute period, followed within 1 hour by continuous IV infusion of 180 mg APL-9 in 250 mL saline at the rate of 15 mg/hour until Day 7 or resolution of ARDS (partial pressure of oxygen [PaO2]/fraction of inspired oxygen [FiO2] ratio >300 millimeter [mm] of mercury [Hg]), whichever occurred earlier. In addition, subjects received institutional SoC to treat their conditions.
- Part 2: APL-9: Subjects received an initial IV infusion of 180 mg APL-9 in 50 mL of saline once over a 10-minute period, followed within 1 hour by continuous IV infusion of 180 mg APL-9 in 250 mL saline at the rate of 15 mg/hour until Day 7 or up to and including Day 21, discontinuation of respiratory support (supplemental oxygen or mechanical ventilation), or hospital discharge, whichever occurred latest. In addition, subjects received institutional SoC to treat their conditions.
- Part 2: Control: Subjects received an initial IV infusion of 50 mL of saline once over a 10-minute period, followed within 1 hour by continuous IV infusion of 250 mL saline at the rate of 21 mL/hour until Day 7 or up to and including Day 21, discontinuation of respiratory support (supplemental oxygen or mechanical ventilation), or hospital discharge, whichever occurred latest. In addition, subjects received institutional SoC to treat their conditions.
Period: Overall Study
Arm/Group | Part 1: APL-9 | Part 2: APL-9 | Part 2: Control
Started | 6 | 34 | 32
Received Treatment | 6 | 33 | 32
Completed (Completed the study) | 5 | 18 | 21
Not Completed | 1 | 16 | 11
Not completed — Death | 1 | 12 | 7
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Sponsor Request | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all subjects who received at least 1 dose of study drug. Subjects were analyzed according to the actual treatment they received.
Groups:
- Part 1: APL-9: Subjects received an initial IV infusion of 180 mg APL-9 in 50 mL of saline once over a 10-minute period, followed within 1 hour by continuous IV infusion of 180 mg APL-9 in 250 mL saline at the rate of 15 mg/hour until Day 7 or resolution of ARDS (PaO2/FiO2 ratio >300 mm Hg), whichever occurred earlier. In addition, subjects received institutional SoC to treat their conditions.
- Total: Total of all reporting groups
Arm/Group | Part 1: APL-9 | Part 2: APL-9 | Part 2: Control | Total
Number analyzed (Participants) | 6 | 33 | 32 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 15 | 18 | 39
  >=65 years | 0 | 18 | 14 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 17 | 13 | 33
  Male | 3 | 16 | 19 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 11 | 12 | 25
  Not Hispanic or Latino | 4 | 13 | 14 | 31
  Unknown or Not Reported | 0 | 9 | 6 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Black/African American | 3 | 3 | 2 | 8
  Native Hawaiian/Pacific Islander | 0 | 0 | 0 | 0
  White | 1 | 21 | 18 | 40
  Unknown or Not Reported | 0 | 4 | 2 | 6
  Unspecified | 2 | 4 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Experienced Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: TEAEs were defined as those adverse events that developed or worsened in severity after initiation of the first dose of study drug and up to 30 (+7) days beyond the last dose of study drug. A serious TEAE was any TEAE or suspected adverse reaction that, in the view of either the Investigator or Sponsor, resulted in any of the following outcomes: death; is life threatening; inpatient hospitalization or prolongation of existing hospitalization; a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; or a congenital anomaly/birth defect.
Time Frame: From the first dose of study drug and up to 30 (+7) days after the last dose of study drug. Part 1: Day 1 up to Day 44; Part 2: Day 1 up to Day 58
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: APL-9 | Part 2: APL-9 | Part 2: Control
Number analyzed (Participants) | 6 | 33 | 32
Participants
  TEAEs | 4 | 23 | 22
  Serious TEAEs | 1 | 14 | 15

2. Secondary Outcome: Hospital Length of Stay
Description: Hospital length of stay was defined as randomization date to hospital discharge. For subjects with death of any cause or withdrawal of study participation, hospital length of stay was imputed with the longest hospital length of stay observed in the study. Median hospital length of stay was estimated using the Kaplan-Meier method.
Time Frame: Part 2: Day 1 up to Day 58
Population: The full analysis set (FAS) included all randomized subjects who received at least 1 dose of study drug. The analyses using the FAS were based upon the actual treatment allocated. Analysis was pre-specified in Part 2 only.
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Part 2: APL-9 | Part 2: Control
Number analyzed (Participants) | 32 | 32
days | 21.5 [8.0 to 47.0] | 15.5 [9.0 to 30.0]
Statistical Analysis 1: Comparison: Part 2: APL-9 vs Part 2: Control; P-value was from a 2-sided stratified Log-rank test by the randomization stratification factors (need of mechanical ventilation [yes vs no] and age [<65 years vs ≥65 years]) at 0.1 significant level for evaluation of treatment difference. Hazard ratio was obtained from a Cox regression model with treatment and the randomization stratification factors as fixed factors and 90% confidence interval (CI) was based on the Wald method; Test type: Superiority; p = 0.82, Log Rank; Hazard Ratio (HR) = 0.98, 90% CI 2-sided [0.63 to 1.51]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as randomization date to death of any cause, censored at the last day known to be alive. Median overall survival was estimated using the Kaplan-Meier method.
Time Frame: Part 2: Day 1 up to Day 58 (until the safety follow-up assessment 30 days after last study treatment [+7 days])
Population: The FAS included all randomized subjects who received at least 1 dose of study treatment. The analyses using the FAS were based upon the actual treatment allocated. Analysis was pre-specified in Part 2 only.
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Part 2: APL-9 | Part 2: Control
Number analyzed (Participants) | 32 | 32
days | NA [27.0 to NA] — The upper CI and median were not calculable due to insufficient events. | NA [NA to NA] — The lower and upper CIs and median were not calculable due to insufficient events.
Statistical Analysis 1: Comparison: Part 2: APL-9 vs Part 2: Control; P-value was from a 2-sided stratified Log-rank test by the randomization stratification factors (need of mechanical ventilation [yes vs no] and age [<65 years vs ≥65 years]) at 0.1 significant level for evaluation of treatment difference. Hazard ratio was obtained from a Cox regression model with treatment and the randomization stratification factors as fixed factors and 90% CI was based on the Wald method; Test type: Superiority; p = 0.36, Log Rank; Hazard Ratio (HR) = 1.62, 90% CI 2-sided [0.77 to 3.40]

4. Secondary Outcome: Change From Baseline in Sequential Organ Failure Assessment (SOFA) Score Over Time
Description: The SOFA score is an aggregate score based on objective measures of 6 organ systems: respiratory, coagulation, hepatic, cardiovascular, neurologic, and renal. The minimum value is 0 and maximum value is 24. Higher scores indicate worse outcomes. A subject with a SOFA score of zero was defined as being free of organ failure.
Time Frame: Part 2: Baseline (Day 1) and Days 3, 5, 7, 11, 15 and end of treatment (EOT) visit (up to Day 21)
Population: The FAS included all randomized subjects who received at least 1 dose of study drug. The analyses using the FAS were based upon the actual treatment allocated. Analysis was pre-specified in Part 2 only. Only subjects with values at both Baseline and the specified visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part 2: APL-9 Plus SoC: Subjects received an initial IV infusion of 180 mg APL-9 in 50 mL of saline once over a 10-minute period, followed within 1 hour by continuous IV infusion of 180 mg APL-9 in 250 mL saline at the rate of 15 mg/hour until Day 7 or up to and including Day 21, discontinuation of respiratory support (supplemental oxygen or mechanical ventilation), or hospital discharge, whichever occurred latest. Follow-up safety assessments were collected 30 days following the last dose of study treatment (with a +7-day window). All subjects received SoC independent of their randomization.
- Part 2: Vehicle Control Plus SoC: Subjects received an initial IV infusion of 50 mL of saline once over a 10-minute period, followed within 1 hour by continuous IV infusion of 250 mL saline at the rate of 21 mL/hour until Day 7 or up to and including Day 21, discontinuation of respiratory support (supplemental oxygen or mechanical ventilation), or hospital discharge, whichever occurred latest. Follow-up safety assessments were collected 30 days following the last dose of study treatment (with a +7-day window). All subjects received SoC independent of their randomization.
Arm/Group | Part 2: APL-9 Plus SoC | Part 2: Vehicle Control Plus SoC
Number analyzed (Participants) | 31 | 29
score on a scale
  Change to Day 3: number analyzed (Participants) | 22 | 23
  Change to Day 3 | 0.4 (2.17) | 1.2 (2.06)
  Change to Day 5: number analyzed (Participants) | 19 | 24
  Change to Day 5 | 0.6 (3.00) | 0.6 (2.48)
  Change to Day 7: number analyzed (Participants) | 10 | 14
  Change to Day 7 | 1.8 (3.97) | 0.9 (3.50)
  Change to Day 11: number analyzed (Participants) | 3 | 5
  Change to Day 11 | 1.7 (2.08) | 0.2 (5.97)
  Change to Day 15: number analyzed (Participants) | 2 | 2
  Change to Day 15 | 0.0 (2.83) | -1.0 (2.83)
  Change to EOT: number analyzed (Participants) | 23 | 22
  Change to EOT | 0.2 (3.56) | 0.6 (3.98)

5. Secondary Outcome: Total Duration of Mechanical Ventilation
Description: Total duration of mechanical ventilation was calculated from the randomization date and was defined as days on mechanical ventilation during the study participation. For subjects with death of any cause (or withdrawal of study participation), total duration of mechanical ventilation was imputed with the longest duration observed in the study. Any subject who was not on mechanical ventilation at the randomization date was excluded. Median total duration of mechanical ventilation was estimated using the Kaplan-Meier method.
Time Frame: Part 2: Day 1 up to Day 58
Population: The FAS included all randomized subjects who received at least 1 dose of study drug. The analyses using the FAS were based upon the actual treatment allocated. Analysis was pre-specified in Part 2 only.
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Part 2: APL-9 | Part 2: Control
Number analyzed (Participants) | 32 | 32
days | 47.0 [NA to NA] — The lower and upper CIs were not calculable due to insufficient events. | 8.5 [7.0 to NA] — The upper CI was not calculable due to insufficient events.
Statistical Analysis 1: Comparison: Part 2: APL-9 vs Part 2: Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.03, Log Rank; Hazard Ratio (HR) = 0.09, 90% CI 2-sided [0.01 to 0.51]

6. Secondary Outcome: Total Duration of Oxygen Therapy
Description: Total duration of oxygen therapy was calculated from randomization date and was defined as days on mechanical ventilation or supplemental oxygen during the study participation. For subjects with death of any cause (or withdrawal of study participation), total duration of oxygen therapy was imputed with the longest duration observed in the study. Any subject who was not on mechanical ventilation or supplemental oxygen at the randomization date was excluded. Median total duration of oxygen therapy was estimated using the Kaplan-Meier method.
Time Frame: Part 2: Day 1 up to Day 58
Population: as for outcome 3
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Part 2: APL-9 | Part 2: Control
Number analyzed (Participants) | 32 | 32
days | 9.0 [5.0 to 47.0] | 8.0 [7.0 to NA] — The upper CI was not calculable due to insufficient events.
Statistical Analysis 1: Comparison: Part 2: APL-9 vs Part 2: Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.93, Log Rank; Hazard Ratio (HR) = 1.09, 90% CI 2-sided [0.69 to 1.72]

7. Secondary Outcome: Serum Concentration of APL-9 Over Time
Description: To evaluate pharmacokinetics (PK), blood samples were collected at pre-specified timepoints and serum concentrations of APL-9 were determined. Blood was collected 3 times on Day 1: prior to the initial infusion, as soon as possible following the initial infusion (within 5-10 minutes) prior to the continuous infusion, and at 2 hours after the beginning of the continuous infusion. Blood was then collected once daily between 1-2 hours after the first dose on Days 3, 5, 7, 11 (if treatment was ongoing), Day 15 (if treatment was ongoing) and at the EOT visit.
Time Frame: Part 1: Day 1 (pre- and post-dose) and Days 3, 5 and 7 (including EOT visit); Part 2: Day 1 (pre- and post-dose) and Days 3, 5, 7, 11, 15 and EOT visit (up to Day 21)
Population: The PK set included all subjects in the safety set and for whom at least 1 PK sample was evaluable.
Measure: Mean (Standard Deviation); unit: micrograms (μg)/mL)
Groups:
- Control: Subjects received an initial IV infusion of 50 mL of saline once over a 10-minute period, followed within 1 hour by continuous IV infusion of 250 mL saline at the rate of 21 mL/hour until Day 7 or up to and including Day 21, discontinuation of respiratory support (supplemental oxygen or mechanical ventilation), or hospital discharge, whichever occurred latest. In addition, subjects received institutional SoC to treat their conditions.
Arm/Group | Part 1: APL-9 | Part 2: APL-9 | Control
Number analyzed (Participants) | 6 | 33 | 31
micrograms (μg)/mL)
  Day 1, Pre-dose: number analyzed (Participants) | 6 | 30 | 30
  Day 1, Pre-dose | 0.0 (0.00) | 3.9 (11.72) | 0.0 (0.00)
  Day 1, 10 mins: number analyzed (Participants) | 6 | 29 | 30
  Day 1, 10 mins | 48.1 (14.00) | 77.7 (168.78) | 2.6 (13.99)
  Day 1, 2 hours: number analyzed (Participants) | 6 | 26 | 30
  Day 1, 2 hours | 56.2 (14.21) | 54.1 (17.28) | 2.2 (12.00)
  Day 3: number analyzed (Participants) | 6 | 23 | 25
  Day 3 | 98.0 (11.03) | 87.7 (31.87) | 5.0 (24.80)
  Day 5: number analyzed (Participants) | 6 | 18 | 21
  Day 5 | 111.5 (8.14) | 103.7 (21.95) | 2.3 (10.43)
  Day 7: number analyzed (Participants) | 2 | 11 | 13
  Day 7 | 116.0 (2.83) | 121.6 (28.71) | 2.3 (8.32)
  Day 11: number analyzed (Participants) | 0 | 3 | 5
  Day 11 |  | 115.3 (24.54) | 2.6 (5.72)
  Day 15: number analyzed (Participants) | 0 | 2 | 2
  Day 15 |  | 133.4 (60.25) | 2.4 (3.45)
  EOT: number analyzed (Participants) | 3 | 21 | 20
  EOT | 114.5 (16.21) | 95.0 (34.19) | 0.0 (0.00)

8. Secondary Outcome: Change From Baseline at EOT Visit in Biomarkers of Complement Activation: Components C3 and C4
Description: To evaluate pharmacodynamic (PD) parameters, blood samples were collected at pre-specified timepoints. Results are presented for change from baseline to EOT visit for complement biomarkers C3 and C4.
Time Frame: Part 1: Baseline (Day 1) and EOT visit (up to Day 7); Part 2: Baseline (Day 1) and EOT visit (up to Day 21)
Population: The PD set included all subjects in the safety set with at least 1 PD evaluation. Only subjects with values at both Baseline and the EOT visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/deciliter (dL)
Arm/Group | Part 1: APL-9 | Part 2: APL-9 | Part 2: Control
Number analyzed (Participants) | 4 | 14 | 18
mg/deciliter (dL)
  C3 | 38.0 (11.17) | 91.4 (64.00) | 2.1 (35.32)
  C4 | 2.0 (19.30) | -3.9 (16.34) | 0.2 (15.40)

9. Secondary Outcome: Change From Baseline at EOT Visit in Biomarkers of Complement Activation: Components C3a, C4a, C5a and Terminal Complement Complex (TCC)
Description: To evaluate PD parameters, blood samples were collected at pre-specified timepoints. Results are presented for change from baseline to EOT visit for complement biomarkers C3a, C4a, C5a and TCC.
Time Frame: Part 1: Baseline (Day 1) and EOT visit (up to Day 7); Part 2: Baseline (Day 1) and EOT visit (up to Day 21)
Population: The PD set included all subjects in the safety set with at least 1 PD evaluation. Note: C5a was only measured in Part 2 because this biomarker was added in APL9-COV-201 Protocol Amendment 2 which was after the last subject in Part 1 finished the last study dose. Only subjects with values at both Baseline and the EOT visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/mL
Arm/Group | Part 1: APL-9 | Part 2: APL-9 | Part 2: Control
Number analyzed (Participants) | 3 | 19 | 19
nanograms (ng)/mL
  C3a | -69.6 (16.35) | -357.6 (785.69) | -4.0 (240.70)
  C4a | -337.7 (371.70) | -1560.8 (4821.35) | -87.0 (1028.77)
  C5a: number analyzed (Participants) | 0 | 19 | 19
  C5a |  | -6.9 (14.88) | -3.9 (9.77)
  TCC | -143.1 (87.41) | -127.4 (121.90) | -12.2 (337.02)

10. Secondary Outcome: Change From Baseline at EOT Visit in Biomarkers of Complement Activation: Complement Bb
Description: To evaluate PD parameters, blood samples were collected at pre-specified timepoints. Results are presented for change from baseline to EOT visit for complement biomarker Bb, a marker of alternative pathway activation.
Time Frame: Part 1: Baseline (Day 1) and EOT visit (up to Day 7); Part 2: Baseline (Day 1) and EOT visit (up to Day 21)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Part 1: APL-9 | Part 2: APL-9 | Part 2: Control
Number analyzed (Participants) | 3 | 19 | 19
μg/mL | -0.6 (0.13) | -0.9 (0.74) | -0.1 (1.56)

11. Secondary Outcome: Change From Baseline at EOT Visit in Biomarkers of Complement Activation: Alternative Complement Pathway Hemolytic Activity (AH50)
Description: To evaluate PD parameters, blood samples were collected at pre-specified timepoints. Results are presented for change from baseline to EOT visit for complement biomarker AH50.
Time Frame: Part 1: Baseline (Day 1) and EOT visit (Day 7); Part 2: Baseline (Day 1) and EOT visit (up to Day 21)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units (U)/mL
Arm/Group | Part 1: APL-9 | Part 2: APL-9 | Part 2: Control
Number analyzed (Participants) | 3 | 19 | 18
Units (U)/mL | -157.7 (26.84) | -84.3 (44.51) | -2.3 (43.72)

12. Secondary Outcome: Change From Baseline at EOT Visit in Biomarkers of Coagulopathy: Reticulocytes
Description: To evaluate PD parameters, blood samples were collected at pre-specified timepoints. Results are presented for change from baseline to EOT visit for the coagulation biomarker reticulocytes. Percentage (%) of reticulocytes was calculated as (Number of Reticulocytes / Number of Red Blood Cells) X 100.
Time Frame: Part 1: Baseline (Day 1) and EOT visit (Day 7); Part 2: Baseline (Day 1) and EOT visit (up to Day 21)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: % of reticulocytes
Arm/Group | Part 1: APL-9 | Part 2: APL-9 | Part 2: Control
Number analyzed (Participants) | 0 | 4 | 7
% of reticulocytes |  | 10325.4 (20649.77) | 23929.1 (87585.96)

13. Secondary Outcome: Change From Baseline at EOT Visit in Biomarkers of Coagulopathy: Schistocytes
Description: To evaluate PD parameters, blood samples were collected at pre-specified timepoints. Results are presented for change from baseline to EOT visit for the coagulation biomarker schistocytes.
Time Frame: Part 1: Baseline (Day 1) and EOT visit (Day 7); Part 2: Baseline (Day 1) and EOT visit (up to Day 21)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter (L)
Arm/Group | Part 1: APL-9 | Part 2: APL-9 | Part 2: Control
Number analyzed (Participants) | 0 | 0 | 1
10^9 cells/liter (L) |  |  | 0.0 (NA) — Standard deviation was not calculated due to only 1 subject analyzed

14. Secondary Outcome: Change From Baseline at EOT Visit in Biomarkers of Coagulopathy: Lactate Dehydrogenase
Description: To evaluate PD parameters, blood samples were collected at pre-specified timepoints. Results are presented for change from baseline to EOT visit for the coagulation biomarker lactate dehydrogenase.
Time Frame: Part 1: Baseline (Day 1) and EOT visit (Day 7); Part 2: Baseline (Day 1) and EOT visit (up to Day 21)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part 1: APL-9 | Part 2: APL-9 | Part 2: Control
Number analyzed (Participants) | 5 | 16 | 23
U/L | -464.6 (427.86) | -135.2 (186.90) | -106.1 (205.59)

15. Secondary Outcome: Change From Baseline at EOT Visit in Biomarkers of Coagulopathy: D-Dimer and Ferritin
Description: To evaluate PD parameters, blood samples were collected at pre-specified timepoints. Results are presented for change from baseline to EOT visit for the coagulation biomarkers D-dimer and ferritin.
Time Frame: Part 1: Baseline (Day 1) and EOT visit (Day 7); Part 2: Baseline (Day 1) and EOT visit (up to Day 21)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: APL-9 | Part 2: APL-9 | Part 2: Control
Number analyzed (Participants) | 5 | 17 | 24
ng/mL
  D-dimer: number analyzed (Participants) | 4 | 17 | 23
  D-dimer | -783.8 (607.57) | 217.2 (1218.54) | 907.9 (2986.71)
  Ferritin | -133.6 (80.80) | -53.1 (650.97) | -19.3 (694.52)

16. Secondary Outcome: Change From Baseline at EOT Visit in Biomarkers of Coagulopathy: Haptoglobin and Fibrinogen
Description: To evaluate PD parameters, blood samples were collected at pre-specified timepoints. Results are presented for change from baseline to EOT visit for the coagulation biomarkers haptoglobin and fibrinogen.
Time Frame: Part 1: Baseline (Day 1) and EOT visit (Day 7); Part 2: Baseline (Day 1) and EOT visit (up to Day 21)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1: APL-9 | Part 2: APL-9 | Part 2: Control
Number analyzed (Participants) | 4 | 14 | 22
mg/dL
  Haptoglobin: number analyzed (Participants) | 0 | 7 | 14
  Haptoglobin |  | -5435.4 (7571.18) | -4554.0 (7756.60)
  Fibrinogen | -147.3 (170.55) | 3995.1 (15113.49) | -1348.2 (9726.66)

17. Secondary Outcome: Change From Baseline at EOT Visit in Biomarkers of Inflammation: C-reactive Protein (CRP)
Description: To evaluate PD parameters, blood samples were collected at pre-specified timepoints. Results are presented for change from baseline to EOT visit for the inflammatory cytokine CRP.
Time Frame: Part 1: Baseline (Day 1) and EOT visit (Day 7); Part 2: Baseline (Day 1) and EOT visit (up to Day 21)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1: APL-9 | Part 2: APL-9 | Part 2: Control
Number analyzed (Participants) | 4 | 17 | 24
mg/dL | -7.0 (8.67) | 6.4 (41.21) | -3.1 (18.52)

18. Secondary Outcome: Change From Baseline at EOT Visit in Biomarkers of Inflammation: Tumor Necrosis Factor Alpha (TNFα), Interleukin-1-beta (IL-1β) and Interleukin-6 (IL-6)
Description: To evaluate PD parameters, blood samples were collected at pre-specified timepoints. Results are presented for change from baseline to EOT visit for the inflammatory cytokines TNFα, IL-1β and IL-6.
Time Frame: Part 1: Baseline (Day 1) and EOT visit (Day 7); Part 2: Baseline (Day 1) and EOT visit (up to Day 21)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Part 1: APL-9 | Part 2: APL-9 | Part 2: Control
Number analyzed (Participants) | 0 | 19 | 19
picograms/mL
  TNFα |  | 19.6 (62.24) | 10.4 (73.92)
  IL-1β |  | -0.6 (7.15) | -8.1 (22.37)
  IL-6 |  | 203.6 (602.54) | 71.3 (499.84)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug and up to 30 (+7) days after the last dose of study drug. Part 1: Day 1 up to Day 44; Part 2: Day 1 up to Day 58.
Description: The safety set included all subjects who received at least 1 dose of study drug. Subjects were analyzed according to the actual treatment they received.
Arm/Group | Part 1: APL-9 | Part 2: APL-9 | Part 2: Control
All-Cause Mortality (participants affected / at risk) | 1/6 | 13/33 | 8/32
Serious Adverse Events (participants affected / at risk) | 1/6 | 14/33 | 15/32
Other Adverse Events (participants affected / at risk) | 3/6 | 20/33 | 20/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: APL-9 (N=6) | Part 2: APL-9 (N=33) | Part 2: Control (N=32)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 4 | 1
Sepsis (Infections and infestations) | 0 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 2 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0
Cardiac valve vegetation (Infections and infestations) | 0 | 0 | 1
Fungaemia (Infections and infestations) | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1 | 0
Distributive shock (Vascular disorders) | 0 | 1 | 1
Embolism venous (Vascular disorders) | 0 | 1 | 1
Shock (Vascular disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 1
Right ventricular dilatation (Cardiac disorders) | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Blood pH decreased (Investigations) | 0 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: APL-9 (N=6) | Part 2: APL-9 (N=33) | Part 2: Control (N=32)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Lice infestation (Infections and infestations) | 0 | 0 | 1
Nosocomial infection (Infections and infestations) | 0 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 1
Renal failure (Renal and urinary disorders) | 0 | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 1 | 0
Distributive shock (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 3 | 0
Shock (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 1
Poor peripheral circulation (Vascular disorders) | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 3
Bradycardia (Cardiac disorders) | 0 | 2 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 2 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 1
Fibrin D dimer increased (Investigations) | 0 | 1 | 1
Serum ferritin increased (Investigations) | 0 | 0 | 2
Anion gap increased (Investigations) | 0 | 1 | 0
Antibiotic level below therapeutic (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood pH increased (Investigations) | 0 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0
Blood sodium increased (Investigations) | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 1
Brain natriuretic peptide increased (Investigations) | 0 | 1 | 0
Drug trough level (Investigations) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 1 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1 | 0
Monocyte count increased (Investigations) | 0 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 0
Platelet count increased (Investigations) | 0 | 1 | 0
Procalcitonin increased (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Calcium deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 3
Catheter site pain (General disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 2
Agitation (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT04402060/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT04402060/SAP_001.pdf